CLINICAL TRIAL: NCT06357429
Title: Evaluation of the Effect of Cold Application on the LI4 Point After Surgery on Acute Pain, Nausea and Anxiety Level
Brief Title: Evaluation of the Effect of the LI4 Cold Application
Acronym: LI4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ayşegül Alioğulları, PHD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 171002100
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Pain; Nausea; Anxiety
Keywords: postoperative pain; cold application; LI4; anxiety; nausea; after surgical
MeSH Terms: conditions — Pain; Nausea; Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold application (Experimental): The first group consists of the experimental group in which cold application is planned to be applied to the hand LI4 point after surgical intervention
  Interventions: Other: Cold Application
- Control (Experimental): The control group in which routine interventions in the clinic are applied.
  Interventions: Other: Cold Application

INTERVENTIONS:
Other: Cold Application — Cold application was applied to the LI4 acupressure point on the patients' hands using an ice battery.

SUMMARY:
It is an experimental study conducted to evaluate the effectiveness of cold application to the LI4 point of the hand to reduce/eliminate pain, nausea and anxiety in postoperative patients. The population of the study consisted of 116 individuals who underwent abdominal surgery with the open surgery method in a state hospital between February 2022 and November 2022 and were followed up in the inpatient ward. The study was completed with 80 individuals constituting the experimental group (n=40) and the control group (n=40). Patient information form, Mcgill Melzack short pain form, Visual Analog Scale, STAI - TX and Cold Application Evaluation Form were used to collect data. Patients in the experimental group underwent cold application with ice cubes for a total of 20 minutes as 2 minutes of cold application and 15 seconds of waiting 4-6 hours after the patient was admitted to the clinic after surgical intervention. Follow-up was performed before cold application, immediately after cold application, 30 minutes after the end of cold application, 1 hour and 2 hours after the end of cold application.

DETAILED DESCRIPTION:
It is a prospective study in which cold application is planned to reduce/eliminate the pain, nausea and anxiety experienced by patients after surgery. There are 2 different sample groups in the study. The first group consists of the experimental group in which cold application is planned to be applied to the hand LI4 point after surgical intervention and the control group in which routine interventions in the clinic are applied.

Hypotheses H1 The pain levels of individuals who received cold application to the LI4 point after surgery are lower than those who received routine care.

H2 Anxiety levels of individuals who underwent cold application to the LI4 point after surgery are lower than those who received routine care.

H3 The nausea levels of individuals who underwent cold application to the LI4 point after surgery are lower than those who received routine care.

Variables of the Study Independent Variables: Cold Application Dependent Variables: Socio-demographic characteristics, pain level, anxiety level, vital signs (body temperature, blood pressure, pulse, respiration), analgesic drug use, nausea level. The study was conducted in the inpatient wards of a state hospital.

Research data were collected every weekday between February 28, 2022 and November 18, 2022 on Monday-Tuesday-Wednesday-Thursday-Thursday-Friday.

The study population consisted of 116 individuals who underwent abdominal surgery and were followed up in the inpatient ward. Inclusion Criteria

* Over 18 years of age
* Can speak and understand Turkish
* Does not have any cognitive, affective and verbal problems that prevent them from communicating,
* No postoperative complications developed,
* Underwent surgery with general anesthesia,
* No cold allergies,
* Standardized analgesia protocol implemented,
* Intensive care follow-up continues as of the fourth hour of the postoperative period,
* Women without a physical hand or arm disability will be included. Patient information form, Mcgill Melzack short pain form, Visual Analog Scale, STAI - TX and Cold Application Evaluation Form were used to collect data. In order to evaluate the comprehensibility of the forms created for data collection and the designed cold application process, a pre-application was performed with the participation of 10 patients who underwent open surgical intervention in the abdominal region in the inpatient ward of the hospital.

The data of the patients within the scope of the preliminary application were not included in the sample.

After the patient was taken to the individual room, his/her clinical status was evaluated. The purpose of the study, LI4 cold application method and its effect on pain were explained. Life findings were measured. Then, pain assessment was performed using the SCS and Mcgill Pain Scale Short Form. State Anxiety Scale and Trait Anxiety Scale were completed by the researcher using face-to-face interview method. After the end of the application, the patient's vital signs were evaluated. The efficacy of cold application was evaluated with SCS, Mcgill Pain Scale Short Form, State Anxiety Scale. At 30, 60 and 120 minutes after cold application, the same evaluations made after the application were repeated and recorded. After the 120th minute evaluation, the "Cold Application Evaluation Form" was completed.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and understand Turkish
* Does not have any cognitive, affective and verbal problems that prevent them from communicating,
* No postoperative complications (bleeding, infection, etc.),
* Underwent surgery with general anesthesia,
* Standardized analgesia protocol implemented,
* Women without a physical hand or arm disability will be included.

Exclusion Criteria:

* Those with chronic diseases such as diabetes, blood pressure, etc,
* Allergic to cold,
* Women with a certain period of intensive care (excluding postoperative care room) follow-up after surgery will not be included in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Pain Level | 9 Months
  Visual Analog Scale - There are numbers from 0 to 10 on the scale consisting of a 10 cm line used horizontally or vertically. The lowest number on the scale, 0, means "No Pain", 1-4 means "Mild Pain", 5-6 means "Moderate Pain" and 7-10 means "Intolerable Pain".
Nausea Level | 9 Months
  Visual Analog Scale - There are numbers from 0 to 10 on the scale consisting of a 10 cm line used horizontally or vertically. The lowest number on the scale, 0, indicates "No Nausea", 1-4 indicates "Mild Nausea", 5-6 indicates "Moderate Nausea" and 7-10 indicates "Intolerable Nausea".
Anxiety Level | 9 Months
  In the State Anxiety Scale, the answer options collected in four classes are (1) Never, (2) A little, (3) A lot and (4) Completely; the options in the Trait Anxiety Scale are (1) Almost never, (2) Sometimes, (3) Very often and (4) Almost always. There are two types of statements in the scales. These are (1) direct or straight statements and (2) reverse statements. Direct statements express negative emotions, while reversed statements express positive emotions. In direct statements, answers with a value of 4 indicate that anxiety is high. In reversed statements, answers with a value of 1 indicate high anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 on the state anxiety scale and items 21, 26, 27, 30, 33, 36 and 39 on the trait anxiety scale are inverted statements. The total score of both scales ranges between 20-80. An increase in the score indicates an increase in the level of anxiety.
Sensory characteristics, intensity and impact of pain | 9 Months
  The McGill Pain Scale Short Form consists of three parts. Section One: This section includes 15 descriptive word groups. Of these, 11 assess the sensory and 4 assess the perceptual dimension of pain. These descriptive words are rated on an intensity scale from 0 to 3 (0= none, 1= mild, 2= moderate, 3= severe). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. The sensory pain score was 0-33, the perceptual pain score was 0-12, and the total pain score was 0-45. An increase in the score indicates an increase in pain.
  Second Part: In the second part of the form, five word groups ranging from "mild pain" to "unbearable pain" were included to determine the severity of the patient's pain.
  Third Section: In the third part, the patient's current pain intensity was assessed using a visual comparison scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül ALİOĞULLARI, PhD Student, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No